CLINICAL TRIAL: NCT00182351
Title: Evaluation of the Safety, Efficacy and Cost-Effectiveness of Two Strategies for the Diagnosis of Deep Vein Thrombosis
Brief Title: D-Dimer Vs Serial Compression Ultrasound Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Health Canada (Other Government)
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CTMG-1995-DDCUS
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2006-09-08 (Estimated); Status verified 2006-09

CONDITIONS: Deep Vein Thrombosis
Keywords: deep vein thrombosis; d-dimer; serial compression ultrasound
MeSH Terms: conditions — Venous Thrombosis | interventions — fibrin fragment D

INTERVENTIONS:
Procedure: D-dimer
Procedure: Serial Compression Ultrasound

SUMMARY:
To determine whether d-dimer testing can be used to simplify and reduce the costs of the diagnostic approach to patients with clinically suspected deep vein thrombosis

ELIGIBILITY:
Inclusion Criteria:

* first suspected deep vein thrombosis
* no previous venous thromboembolism
* referred to thromboembolism outpatient clinic

Exclusion Criteria:

* comorbid condition limiting survival to less than six months
* contraindication to venography (contrast allergy, etc.)
* receiving long term warfarin therapy
* receiving full dose heparin therapy for more than 48 hours
* absence of symptoms during the five days immediately prior to presentation
* symptoms of pulmonary embolism
* pregnancy
* geographic inaccessibility which precludes follow-up

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 810
Dates: Start 1996-04; Study Completion 1999-07

PRIMARY OUTCOMES:
safety of withholding anticoagulants

SECONDARY OUTCOMES:
deep vein thrombosis
pulmonary embolism
death

CONTACTS AND LOCATIONS:
Overall Officials: Clive Kearon, MB, Study Chair — Hamilton Health Sciences and McMaster University
Locations (3):
- Canada (3):
  - Hamilton Health Sciences - Hamilton General Hospital, Hamilton, Ontario
  - St. Joseph's Hospital, Hamilton, Ontario
  - Hamilton Health Sciences - Henderson Hospital, Hamilton, Ontario

REFERENCES:
- [Result] Kearon C, Ginsberg JS, Douketis J, Crowther MA, Turpie AG, Bates SM, Lee A, Brill-Edwards P, Finch T, Gent M. A randomized trial of diagnostic strategies after normal proximal vein ultrasonography for suspected deep venous thrombosis: D-dimer testing compared with repeated ultrasonography. Ann Intern Med. 2005 Apr 5;142(7):490-6. doi: 10.7326/0003-4819-142-7-200504050-00007. PMID 15809460